CLINICAL TRIAL: NCT04243954
Title: Hydromorphone PCA Intravenously vs Sustained-Release Morphine Orally in Cancer Patients With Severe Pain After Successful Titration: A Multicenter, Randomized, Controlled, Phase II Trial
Brief Title: Intravenous vs Oral Analgesia in Cancer Patients With Severe Pain After Successful Titration
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMORCT09-2
Record Dates: First submitted 2020-01-10; First posted 2020-01-28 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-02

CONDITIONS: Cancer Pain
Keywords: Orally; PCA intravenously; Analgesia; Severe cancer pain
MeSH Terms: conditions — Cancer Pain; Agnosia | interventions — Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PCA IV Hydromorphone (continuous dose = 0) (Experimental): 1. Intravenous PCA with hydromorphone after successful titration of 24 hours.
  2. The PCA setting:
  1) Continuous dose = 0; 2) Bolus dose = 10-20% of the total dosage of hydromorphone in the previous 24 hours: 3) Lockout time = 10 minutes; 4) Evaluate once every 24 hours
  Interventions: Drug: PCA IV Hydromorphone (continuous dose = 0)
- PCA IV Hydromorphone (continuous dose ≠ 0) (Experimental): 1. Intravenous PCA with hydromorphone after successful titration of 24 hours.
  2. The PCA setting:
  1) Continuous dose (dose/hours) = the total dosage of hydromorphone in the previous 24 hours/24; 2) Bolus dose = 10-20% of the total dosage of hydromorphone in the previous 24 hours; 3) Lockout time = 10 minutes; 4) Evaluate once every 24 hours
  Interventions: Drug: PCA IV Hydromorphone (continuous dose ≠ 0)
- Oral Morphine (Active Comparator): 1. Swift to sustained-release morphine orally as background dose with immediate release morphine orally for breakthrough pain after successful titration of 24 hours.
  2. Administration of morphine orally 1) Sustained-release morphine orally (dose/12 hours) = the total equianalgesic of the previous 24 hours/2×75% for d1; the total equianalgesic of the previous 24 hours/2 for day 2 and day 3; 2) Immediate release morphine orally = 10-20% of the total equianalgesic of the previous 24 hours; 3) Evaluate once every 24 hours
  Interventions: Drug: Oral morphine

INTERVENTIONS:
Drug: PCA IV Hydromorphone (continuous dose = 0) — Intravenous PCA with hydromorphone after successful titration of 24 hours. the PCA setting: 1) continuous dose = 0; 2) bolus dose = 10-20% of the total dosage of hydromorphone in the previous 24 hours: 3) lockout time = 10 minutes; 4) evaluate once every 24 hours
  Arms: PCA IV Hydromorphone (continuous dose = 0)
Drug: PCA IV Hydromorphone (continuous dose ≠ 0) — Intravenous PCA with hydromorphone after successful titration of 24 hours. the PCA setting: 1) continuous dose (dose/hours) = the total dosage of hydromorphone in the previous 24 hours/24; 2) bolus dose = 10-20% of the total dosage of hydromorphone in the previous 24 hours; 3) lockout time = 10 minutes; 4) evaluate once every 24 hours
  Arms: PCA IV Hydromorphone (continuous dose ≠ 0)
Drug: Oral morphine — Swift to sustained-release morphine orally as background dose with immediate release morphine orally for breakthrough pain after successful titration of 24 hours.
  Administration of morphine orally 1) Sustained-release morphine orally (dose/12 hours) = the total equianalgesic of the previous 24 hours/2×75% for d1; the total equianalgesic of the previous 24 hours/2 for day 2 and day 3; 2) Immediate release morphine orally = 10-20% of the total equianalgesic of the previous 24 hours; 3) Evaluate once every 24 hours
  Arms: Oral Morphine

SUMMARY:
Pain is one of the most common and fear symptoms for cancer patients, which seriously affects the quality of life in cancer patients. At present, oral opioid is the most common route to administrate cancer pain. However, the patients do not satisfy the pain administration with oral opioid after successful titration in many cases, especially the cases with severe cancer pain. Patient controlled analgesia (PCA) with hydromorphone can take analgesic effect rapidly. The aim of this trial is to compare the maintenance with hydromorphone PCA intravenously or switch to Sustained-Release Morphine orally after successful titraton with hydromorphone PCA intravenously in severe cancer pain.

ELIGIBILITY:
Inclusion Criteria:

1. The patients were 18-80 years old and diagnosed as malignant tumor by pathology;
2. Patients with cancer pain is NRS pain score ≥ 7 during previous 24 hours;
3. Patients who will not be treated with radiotherapy within 7 days prior to randomization and during study ;
4. Patients who need chemotherapy, long term administration of hormone, targeted therapy, or bisphosphonates therapy should undergo a stable anti- tumor therapy prior to randomization ;
5. Patients or his/her caregivers who are able to fill out the questionnaire forms ;
6. Ability to correctly understand and cooperate with medication guidance of doctors and nurses ;
7. Without psychiatric problems;
8. ECOG performance status ≤3;
9. Not participated in another drug clinical trial within one month before inclusion（including hydromorphone）;
10. The subjects voluntarily signed the informed consent.

Exclusion Criteria:

1. The pain is confirmed not due to cancer;
2. Patients with severe post-operative pain;
3. Patients with paralytic ileus;
4. Patients with brain metastasis;
5. Patients hypersensitive to opioids;
6. Patients with abnormal lab results that have obvious clinical significance, such as creatine ≥ 2 fold of upper limit of normal value, alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 2.5 fold of upper limit of normal value, or liver function of Child C grade;
7. Patients who cannot take drugs orally;
8. Patients with an incoercible nausea or vomiting;
9. Those who have received monoamine oxidase inhibitor (MAOI) within two weeks before randomization;
10. Patients who are pregnant or in lactation, or who plan to be pregnant within one month after the trial;
11. Those with opioid addiction;
12. Alcoholic patients;
13. Those with cognitive dysfunction;
14. Those with severe depression;
15. Patients with other conditions or reasons causing the patients unable to complete the clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2020-04-10 (Actual); Primary Completion 2020-10-21 (Actual); Study Completion 2020-11-21 (Actual)

PRIMARY OUTCOMES:
Mean pain score | From day1 to day3
  The Numerical Rating Scale (NRS, a score of 0 means no pain and 10 means the most severe) is used to assess the severity of pain. NRS of 24 hours is assessed every day. The mean pain score is a sum of NRS of day 1 (the day after successful titration of 24 hours) to day 3 divided by 3.
  If the NRS of the morphine orally group >3, the NRS in the hydromorphone PCA intravenously group declines more than 30% compared to morphine orally group, which is regards a positive result.
Number of Breakthrough cancer Pain (BTcP) episodes | From day1 to day3
  If NRS of the morphine orally group pain score ≤3 , or if NRS in the hydromorphone PCA intravenously group declines less than 30% compared to morphine orally group, number of Breakthrough cancer Pain (BTcP) episodes in the one of both the hydromorphone PCA intravenously group declines less than 30% compared to morphine orally group, which is regards a positive result.

SECONDARY OUTCOMES:
Number of patients with an average NRS pain score> 3 | From day1 to day3
  The Numerical Rating Scale (NRS, a score of 0 means no pain and 10 means the most severe) is used to assess the severity of pain.
Number of patients with an average NRS pain score> 6 | From day1 to day3
  The Numerical Rating Scale (NRS, a score of 0 means no pain and 10 means the most severe) is used to assess the severity of pain.
Total dosage of opioids | 3 days
  The total dosage of opioids in day 1 to day 3 (day 1 is the day after successful titration of 24 hours)
Satisfaction score | 3 days
  The satisfaction score of the patients to analgesia was evaluated by 10-point scale: 0 points for dissatisfaction, 10 points for very satisfied, the higher the score, the higher the satisfaction.
Quality of life of patients | At 24 hours
  Chinese version of the Edmonton Symptom Assessment System.
Number of patients who switched/discontinued therapy due to serious adverse events or lack of pain control | 3 days
  The number of patients who switched/discontinued therapy due to serious adverse events or lack of pain control

CONTACTS AND LOCATIONS:
Overall Officials: Rongbo Lin, MD, Principal Investigator — Fujian Cancer Hospital
Locations (1):
- China, Fujian, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No